CLINICAL TRIAL: NCT04932005
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of DZD2269 Oral Tablet Following Single and Multiple Ascending Dose Administration to Healthy Adult Participants
Brief Title: A Study of DZD2269 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DZ2021A0001
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DZD2269 (Experimental): This study includes two parts. In Part A, a single dose of DZD2269 at different dose levels will be given. In Part C, DZD2269 at selected dose levels will be given twice daily for 7 days.
  Interventions: Drug: DZD2269
- Placebo (Placebo Comparator): In Part A, a single oral dose of placebo will be given. In Part C, placebo will be given twice daily for 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DZD2269 — Part A: A single oral dose at 5mg, 10mg, 20mg, 40mg, 80mg, 160mg. Part C: Twice daily dosing for 7 days at 10mg, 30mg, 80mg.
  Arms: DZD2269
Drug: placebo — Part A: A single oral dose. Part C: Twice daily dosing for 7 days.
  Arms: Placebo

SUMMARY:
This is a research study in healthy participants. The purpose of this study is to see how safe the study drug is and how well it is tolerated after dosing. This study will also investigate pharmacokinetics of DZD2269; renal excretion of DZD2269 will also be evaluated. The study will also measure biomarkers such as pCREB in the blood.

DETAILED DESCRIPTION:
A phase 1, randomized, double-blinded, placebo-controlled, study in healthy participants. This study includes two parts, Part A (single ascending dose escalation) and Part C (multiple ascending dose escalation).

ELIGIBILITY:
"Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participants must be able to understand the nature of the trial and provide a signed and dated, written informed consent form prior to any study specific procedures, sampling and analyses.
2. Female and/or male aged 18 ~ 55 years, inclusive. Body mass index (BMI) 18 ~ 30 kg/m2, inclusive. Body weight of ≥ 45 kg (Female) or ≥ 55 kg (Male).
3. Healthy as determined by medical history, physical examination, laboratory parameters, vital signs, ECG and pulmonary function test performed before first administration of the study drug.
4. Adequate organ function including hepatic, renal, cardiac and bone marrow function as determined by the investigator.
5. No nicotine use within 3 months.
6. Female participants must have negative pregnancy tests at screening and check-in AND: have been surgically sterile (with documentation of hysterectomy, bilateral oophorectomy, bilateral salpingectomy, bilateral tubal ligation/tubal occlusion) OR post-menopausal (no menstruation for a minimum of 12 months and confirmed by follicle stimulating hormone (FSH) and serum estradiol at screening) OR, if of child-bearing potential, must be using an acceptable method of contraception such as an intrauterine device (IUD), implant or contraceptive injection, or two forms of the following (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge) for the last three months. All females must agree to continue to use their method of birth control for the duration of the study and for a minimum of one complete menstrual cycle.
7. Male participants must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) during the study (from the time they sign consent) and for 6 months after the last dose of the study drug to prevent pregnancy with a partner.

Participants are excluded from the study if any of the following criteria apply:

1. Reported history or any clinically significant abnormalities at screening of cardiac, hepatic, renal, respiratory, GI, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease. Include but not limited to

   * Reported ongoing or prior pulmonary disease including asthma, chronic obstructive pulmonary disease, interstitial lung disease and pneumonitis including but not limited to drug-related pneumonitis.
   * A reported history of additional risk factors for torsade de pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT syndrome).
   * Mean resting corrected QTcF interval (QTC) > 450 msec on screening triplicate electrocardiogram (ECG).
   * Manifestations of malabsorption due to prior GI surgery, reported GI disease, or for an unknown other reason that may affect the absorption of DZD2269
   * Refractory nausea, vomiting and chronic gastrointestinal diseases
   * Resting blood pressure > 140/90 mmHg at screening (a single repeat measurement is allowed if the initial measurement is outside these limits). Resting pulse rate < 45 beats per minute.
2. Infections including:

   * History of known latent or active tuberculosis (TB), or positive screening results according to local recommendations.
   * Positive Hepatitis B surface antigen (HbsAg) or positive hepatitis C virus (HCV) antibodies or confirmed positive HIV test result.
   * Positive polymerase chain reaction (PCR) testing for COVID-19 at admission to clinic.
   * Bacterial infections including pneumonia within 30 days.
   * Other known active infection at the time of screening.
3. Self-reported substance abuse (eg, alcohol, licit or illicit drugs) within 12 months of screening.
4. Testing positive for alcohol and/or drugs-of-abuse.
5. Has donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months prior to receiving the study drug.
6. History of malignancy of any type, with the exception of the following: surgically excised non-melanomatous skin cancers more than 5 years prior to receiving the study drug.
7. History of severe allergy or hypersensitivity reaction or ongoing allergy or hypersensitivity reaction, as judged by investigator
8. Use of any over-the-counter or prescription medications within 14 days or 5 half-lives (whichever is longer), prior to receiving the study drug.
9. Ingestion of herbal medicines within 3 weeks before screening, and grapefruit, grapefruit juice, pomegranate juice, star fruit or orange marmalade (made with Seville oranges) within 1 week prior to screening.
10. Any major surgery within 4 weeks before study drug administration.
11. Blood transfusion within 4 weeks before the study drug administration.
12. Live vaccination within 4 weeks before the study drug administration.
13. COVID-19 vaccination within 2 weeks before the study drug administration.
14. Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) prior to the first dose of investigational study drug with another investigational medication or current enrolment in another investigational drug or post-marketing study.
15. Involvement in the planning and/or conduct of the study (applies to both Dizal staff and/or staff at the study site).
16. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
17. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
18. Any condition or finding that in the Investigators opinion would put the participant or study conduct at risk if the participant were to participate in the study"

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with adverse event (AE) | From first dose until 5 days after the last dose (Up to 6 days for Part A; 12 days for Part C)
  "To assess the safety and tolerability of DZD2269 versus placebo following oral administration"
Number and percentage of participants with serious adverse event (SAE) | From screening until 5 days after the last dose (Up to 34 days for Part A, 40 days for Part C)
  To assess the safety and tolerability of DZD2269 versus placebo following oral administration
Number and percentage of participants with clinically defined abnormal laboratory values | From screening until 5 days after the last dose (Up to 34 days for Part A, 40 days for Part C)
  To assess the safety and tolerability of DZD2269 versus placebo following oral administration
Number and percentage of participants with clinically defined abnormal vital signs | From screening until 5 days after the last dose (Up to 34 days for Part A, 40 days for Part C)
  To assess the safety and tolerability of DZD2269 versus placebo following oral administration
Number and percentage of participants with clinically defined ECG abnormalities | From screening until 5 days after the last dose (Up to 34 days for Part A, 40 days for Part C)
  To assess the safety and tolerability of DZD2269 versus placebo following oral administration

SECONDARY OUTCOMES:
Drug concentrations of DZD2269 in plasma | After the first dose, 6 days for Part A; 7 days for Part C
  To characterize pharmacokinetics of DZD2269 following oral administration in healthy participants
Maximum plasma concentration (Cmax) of DZD2269 | After the first dose, 6 days for Part A; 7 days for Part C
  To characterize pharmacokinetics of DZD2269 following oral administration in healthy participants
Area under the plasma concentration-time curve (AUC) of DZD2269 | After the first dose, 6 days for Part A; 7days for Part C
  To characterize pharmacokinetics of DZD2269 following oral administration in healthy participants

OTHER OUTCOMES:
Percent of Phosphorylated cAMP (Adenosine 3'5' Cyclic Monophosphate)-Response Element Binding protein (pCREB) inhibition in T cells | After the first dose, 2 days for Part A; 7 days for Part C
  To assess modulation of CREB phosphorylation in T cells (whole blood sample) by DZD2269
Concentration of DZD2269 in urine | On Day 7
  To evaluate DZD2269 excretion via urine following multiple oral dosing in healthy participants (Part C only)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Principal Investigator — Frontage Clinical Services, Inc.; Lisa Diamond, PhD, Study Director — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Service 200 Meadowlands Parkway, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No